CLINICAL TRIAL: NCT01615588
Title: The Glycaemic Index of Manuka Honey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Waiariki Institute of Technology (Other)
Collaborators: Manuka Health New Zealand (Other)
Responsible Party: Principal Investigator, Dr Lynne Chepulis, Senior Lecturer, Waiariki Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Manuka GI Study
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: manuka honey; glycaemic index; blood glucose control; individuals; current disease; medication use

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- honey (Experimental): Manuka honey
  Interventions: Dietary Supplement: Manuka Honey

INTERVENTIONS:
Dietary Supplement: Manuka Honey — honey was weighed out to provide 25 g of available carbohydrate in 200 ml of water
  Other Names: Manuka Health New Zealand Manuka honey

SUMMARY:
Five high methylglyoxal (460-667 mg/kg) Manuka honey samples were selected from different geographical locales around the North Island of New Zealand and tested for glycaemic index (GI) in 10 healthy volunteers in a single-blinded, randomised study. Participants were fed honey containing 25g of available carbohydrate in 200 ml water and the blood glucose responses measured (area under the curve; AUC) and compared to that of 25 g of available carbohydrate from glucose.

ELIGIBILITY:
Inclusion Criteria:

* healthy (Body mass index (BMI) 20-25)
* non-smoking
* aged between 18-45 years
* absence of diabetes or chronic illness
* not taking any medications.

Exclusion Criteria:

* currently dieting
* suffering from illness or chronic disease
* currently taking medication
* smokers (including recreational)
* outside healthy BMI range

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determine the Glycaemic index of Manuka honey | 2 weeks
  10 healthy individuals consumed honey (25g of available carbohydrate in 200 ml of water) in a fasted state. Blood glucose levels were recorded at 0, 15, 30, 45, 60, 90 and 120 mins and the area under the blood glucose curve was calculated. All 10 participants took five different honeys and a glucose standard on six different days (with randomised allocation of samples).

CONTACTS AND LOCATIONS:
Locations (1):
- Waiariki Institute of Technology, Rotorua, BOP, New Zealand